CLINICAL TRIAL: NCT00006183
Title: Hematocrit Strategy in Infant Heart Surgery
Brief Title: Comparison of Hematocrit Levels in Infant Heart Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Jane. W. Newburger, M.D., Principal Investigator, Children's Hospital Boston
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: 131; U01HL063411 (NIH)
Record Dates: First submitted 2000-08-21; First posted 2000-08-22 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2008-03

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Heart Defects, Congenital; Transposition of Great Vessels
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Heart Defects, Congenital; Transposition of Great Vessels | interventions — Cardiopulmonary Bypass; Thoracic Surgical Procedures

INTERVENTIONS:
Procedure: Cardiopulmonary Bypass with Two Different Intra-Operative Hematocrits
Procedure: Thoracic Surgery

SUMMARY:
The purpose of this study is to compare the effects of diluted hematocrit (HCT) levels of 35% versus 25% during hypothermic cardiopulmonary bypass (CPB) in infants with d-transposition of the great arteries, a malformation of the heart vessels.

DETAILED DESCRIPTION:
BACKGROUND:

The optimal degree of hemodilution during profoundly hypothermic CPB remains controversial, and widely dissimilar hemodilution studies have evolved at centers that perform infant cardiac surgery. HCT, a measurement of the volume of red blood cells, is of interest in cardiopulmonary bypass. Higher HCT levels expose individuals to the risks of microvascular occlusion (blockage in the small blood vessels), while lower HCT levels may critically limit oxygen delivery to the brain and other organs. Preliminary research suggests that higher HCT levels provide superior brain and myocardial protection, but there have not been any studies that report on outcomes after usage of higher versus lower HCT levels.

DESIGN NARRATIVE:

In this single-center, prospective, randomized study, hemodilution to a HCT level of 35% versus 25% will be compared with respect to neurodevelopmental outcome and early postoperative course in infants with congenital heart disease. The first aim of this study will test the hypothesis that hemodilution to a HCT level of 35%, compared to a level of 25%, will be associated with superior central nervous system protection. The primary outcome variable will be developmental outcome at age 1 year, assessed using the Bayley Scales of Infant Development. Secondary outcome variables include the following: 1) tissue release of S-100 protein as a measure of cerebral cellular injury; 2) cerebral hemodynamics and oxygenation, determined by near infrared spectroscopy (NIRS); 3) intrinsic cerebral vasoregulation, measured by NIRS and transcranial Doppler; and 4) at age 1 year, neurologic examination, the MacArthur inventory, and structural and volumetric findings of magnetic resonance imaging (MRI).

The second aim of this study will test the hypothesis that hemodilution to a HCT level of 35%, compared to a level of 25%, will be associated with better early postoperative cardiovascular status. The primary outcome measure will be serum lactate levels 1 hour after the surgery. Secondary outcome measures will include the following: 1) the duration of postoperative endotracheal intubation, ICU stay, and hospital stay; 2) serum lactate levels; 3) the PaO2/FiO2 ratio; 4) levels of circulating pro-inflammatory cytokines; and 5) the percent change in total body water, estimated by bioelectrical impedance. The structure of the study will allow assessment of whether 1-year outcomes can be predicted by perioperative variables other than the HCT strategies. Through the use of novel techniques such as NIRS and volumetric MRI, the study may also provide insight into mechanisms by which HCT and other perioperative variables affect the brain. The information obtained from this study should be broadly generalized to infants with other forms of congenital heart disease undergoing early repair and should have substantial impact on clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing repair of ventricular septal defect within 9 months of study entry
* Tetralogy of fallot
* D-transposition of the great arteries
* Atrio-ventricular septal defect

Exclusion Criteria:

* Birth weight less than 2.3 kg
* Recognizable phenotypic syndrome of congenital anomalies
* Extracardiac anomalies of greater than minor severity
* Previous cardiac surgery
* Associated cardiovascular anomalies requiring aortic arch reconstruction or additional open surgical procedures before the planned developmental follow-up

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120
Dates: Start 2000-07; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Serum lactate levels (measured 1 hour after surgery)
Developmental outcome (measured by Bayley Scales of Infant Development at age 1 year)

SECONDARY OUTCOMES:
Duration of postoperative endotracheal intubation, ICU stay, and hospital stay
PaO2/FiO2 ratio
Levels of circulating pro-inflammatory cytokines
Percent change in total body water, as estimated by bioelectrical impedance (measured 1 hour after surgery)
Tissue release of S-100 protein as a measure of cerebral cellular injury
Cerebral hemodynamics and oxygenation, as determined by near infrared spectroscopy (NIRS)
Intrinsic cerebral vasoregulation, as measured by NIRS and transcranial Doppler
Neurologic factors, as determined by neurologic examination, the MacArthur inventory, and structural and volumetric findings of MRI (measured at age 1 year)

CONTACTS AND LOCATIONS:
Overall Officials: Jane W. Newburger, MD, MPH, Study Chair — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Children's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Jonas RA, Wypij D, Roth SJ, Bellinger DC, Visconti KJ, du Plessis AJ, Goodkin H, Laussen PC, Farrell DM, Bartlett J, McGrath E, Rappaport LJ, Bacha EA, Forbess JM, del Nido PJ, Mayer JE Jr, Newburger JW. The influence of hemodilution on outcome after hypothermic cardiopulmonary bypass: results of a randomized trial in infants. J Thorac Cardiovasc Surg. 2003 Dec;126(6):1765-74. doi: 10.1016/j.jtcvs.2003.04.003. PMID 14688685
- [Background] Bassan H, Gauvreau K, Newburger JW, Tsuji M, Limperopoulos C, Soul JS, Walter G, Laussen PC, Jonas RA, du Plessis AJ. Identification of pressure passive cerebral perfusion and its mediators after infant cardiac surgery. Pediatr Res. 2005 Jan;57(1):35-41. doi: 10.1203/01.PDR.0000147576.84092.F9. Epub 2004 Nov 5. PMID 15531739
- [Background] Kussman BD, Wypij D, DiNardo JA, Newburger J, Jonas RA, Bartlett J, McGrath E, Laussen PC. An evaluation of bilateral monitoring of cerebral oxygen saturation during pediatric cardiac surgery. Anesth Analg. 2005 Nov;101(5):1294-1300. doi: 10.1213/01.ANE.0000180205.85490.85. PMID 16243983
- [Derived] Rollins CK, Asaro LA, Akhondi-Asl A, Kussman BD, Rivkin MJ, Bellinger DC, Warfield SK, Wypij D, Newburger JW, Soul JS. White Matter Volume Predicts Language Development in Congenital Heart Disease. J Pediatr. 2017 Feb;181:42-48.e2. doi: 10.1016/j.jpeds.2016.09.070. Epub 2016 Nov 9. PMID 27837950
- [Derived] Kussman BD, Wypij D, Laussen PC, Soul JS, Bellinger DC, DiNardo JA, Robertson R, Pigula FA, Jonas RA, Newburger JW. Relationship of intraoperative cerebral oxygen saturation to neurodevelopmental outcome and brain magnetic resonance imaging at 1 year of age in infants undergoing biventricular repair. Circulation. 2010 Jul 20;122(3):245-54. doi: 10.1161/CIRCULATIONAHA.109.902338. Epub 2010 Jul 6. PMID 20606124
- [Derived] Kipps AK, Wypij D, Thiagarajan RR, Bacha EA, Newburger JW. Blood transfusion is associated with prolonged duration of mechanical ventilation in infants undergoing reparative cardiac surgery. Pediatr Crit Care Med. 2011 Jan;12(1):52-6. doi: 10.1097/PCC.0b013e3181e30d43. PMID 20453699
- [Derived] Soul JS, Robertson RL, Wypij D, Bellinger DC, Visconti KJ, du Plessis AJ, Kussman BD, Scoppettuolo LA, Pigula F, Jonas RA, Newburger JW. Subtle hemorrhagic brain injury is associated with neurodevelopmental impairment in infants with repaired congenital heart disease. J Thorac Cardiovasc Surg. 2009 Aug;138(2):374-81. doi: 10.1016/j.jtcvs.2009.02.027. Epub 2009 Apr 10. PMID 19619781
- [Derived] Newburger JW, Jonas RA, Soul J, Kussman BD, Bellinger DC, Laussen PC, Robertson R, Mayer JE Jr, del Nido PJ, Bacha EA, Forbess JM, Pigula F, Roth SJ, Visconti KJ, du Plessis AJ, Farrell DM, McGrath E, Rappaport LA, Wypij D. Randomized trial of hematocrit 25% versus 35% during hypothermic cardiopulmonary bypass in infant heart surgery. J Thorac Cardiovasc Surg. 2008 Feb;135(2):347-54, 354.e1-4. doi: 10.1016/j.jtcvs.2007.01.051. PMID 18242267